CLINICAL TRIAL: NCT03060564
Title: A Randomized, Prospective Trial Comparing Reconstruction Of Acute Coracoclavicular Ligament Disruption With and Without Tendon Graft
Brief Title: Reconstruction Of Acute Coracoclavicular Ligament Disruption With and Without Tendon Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Brian Lee (Other)
Collaborators: Cedars-Sinai Medical Center (Other); Kerlan-Jobe Institute (Unknown); White Memorial Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Brian Lee, orthopedic surgeon specializing in arthroscopic and open surgery of all conditions of the shoulder and elbow including arthritis, tendon disorders, fractures, and instability, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro46696
Record Dates: First submitted 2017-02-07; First posted 2017-02-23 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Acromioclavicular Joint Dislocation
Keywords: shoulder; orthopaedics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AC repair with tendon graft (Experimental): acromioclavicular repair with tendon graft.
  Interventions: Procedure: tendon graft
- AC repair with no tendon graft (Active Comparator): acromioclavicular repair without tendon graft/no intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Procedure: tendon graft — JRF Orthopedics Tendon Graft
  Arms: AC repair with tendon graft
Other: No intervention — No intervention
  Arms: AC repair with no tendon graft

SUMMARY:
To evaluate patient function, radiographic changes and complication rates of acute coracoclavicular (CC) joint reconstruction with and without the use of tendon graft as an augmentation to repair.

DETAILED DESCRIPTION:
Acromioclavicular (AC) joint dislocations comprise up to 12% of shoulder girdle injuries. Many methods of reconstructing the coracoclavicular ligaments, which provide vertical stability of the acromioclavicular joint, have been described. The use of tendon graft to augment the reconstruction provides improved biomechanical stability, less radiographic changes postoperatively including loss of reduction, and improved function. However, the use of a tendon graft necessitates larger drill holes in the clavicle when compared to suture-only repair constructs. The size and placement of these tunnels in the clavicle have been associated with a higher rate of complications.

It has been shown that repairs in the setting of acute injury demonstrate less complications including loss of reduction when compared with chronic dislocations. However, other reports describing repair of acute AC joint dislocations without graft augmentation have described significant changes in coracoclavicular distance with routine follow up radiographs, and up to 90% implant migration rates. While use of tendon graft would be expected to provide further stability, they may in turn cause an increased complication rate.

1. To determine complication rates in the reconstruction of AC joint dislocations with and without the use of tendon graft.
2. Determine patient satisfaction, the ASES, Constant, SF-12, SANE, SST scores of shoulders that undergo reconstruction of acute AC joint dislocations with and without the use of graft.
3. The investigation aims to determine whether or not graft should be used in the reconstruction of acute AC joint dislocations.

ELIGIBILITY:
Inclusion Criteria:

* Displaced acromioclavicular joint dislocation sustained within 3 weeks of surgery
* recommended for operative fixation
* age 18 years or older

Exclusion Criteria:

* Open dislocation
* previous acromioclavicular surgery
* unable to follow study protocol
* concomitant injury requiring surgery (rotator cuff repair, biceps tenotomy/tenodesis)
* active infection
* unable to follow postoperative rehabilitation guidelines
* reconstruction with coracoclavicular screw or hook plate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Complication Rates with and without the use of graft tendons | 2 years
  loss of radiographic reduction, infection, need for more surgery
(American Shoulder Elbow Society (ASES) | 2 years
  Shoulder Function survey (17 multiple choice questions).
Instability Index Constant Score (ISIS) | 2 years
  Shoulder Instability survey for last 4 weeks (yes/no and multiple choice). Score is graded poor, fair, good, excellent.
Simple Shoulder Test (SST) | 2 years
  Shoulder Function survey (12 yes/no questions)
Short Form-12 | 2 years
  This survey assesses patient's health satisfaction. This information will help keep track of how patients feel and how well patients are able to do your usual activities. (12 multiple choice questions)
Single Assessment Numerical Evaluation (SANE) | 2 years
  Patient assessment rating from 0-100 shoulder normality
Visual Analog Score (VAS) | 2 years
  Measurement of shoulder pain from 0 (no pain) to 10 (unbearable distress)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lee, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Kerlan-Jobe Institute at White Memorial Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No